CLINICAL TRIAL: NCT04412980
Title: Importance of Ionized Magnesium Measurement for Monitoring of Continuous Venovenous Haemodialysis With Citrate Anticoagulation
Brief Title: Ionized Magnesium for Monitoring of Citrate-anticoagulated CVVHD
Acronym: MagiCC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Novamedica Laboratories (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0121
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-05

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Continuous renal replacement therapy with regional citrate anticoagulation (CRRT-RCA); Ionized hypomagnesemia; Monitoring of ionized magnesemia; Morbi-moratlity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been reported in several studies that ionized hypomagnesemia is associated with higher morbidity and mortality rates. During continuous renal replacement therapy with regional citrate anticoagulation (CRRT-RCA), the loss of magnesium has been reported to not be covered by magnesium concentration in ordinary dialysis fluid. This may lead to ionized hypomagnesemia. However the incidence of ionized hypomagnesemia in patients requiring CRRT-RCA remains unclear and need to be estimated to determine if ionized magnesium monitoring could be of interest. This study aim to assess the incidence of ionized hypomagnesemia induced by CRRT-RCA.

ELIGIBILITY:
Inclusion criteria:

* Consecutive patients admitted to the ICU and requiring continuous renal replacement therapy with regional citrate anticoagulation
* age > 18 ans

Exclusion criteria:

* Persons under protection
* Paritcipation rejections

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU and requiring CRRT-RCA
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
assess the systemic ionized magnesemia change after 24h of CRRTsystemic variations of iMg | Day 0 and Day 1
  assess the systemic ionized magnesemia change after 24h of CRRT wiith regional citrate anticoagulation

SECONDARY OUTCOMES:
Proportion of patients with heart rhythm disturbances | 1 day
  Proportion of patients with heart rhythm disturbances
Assessment of morbidity and mortality | 1 day
  Assessment of morbidity and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Romaric Larcher, MD PhD, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC